CLINICAL TRIAL: NCT04907734
Title: Differences in Skinfold Thickness Depending on the Caliper Used.
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Esparza Ros, Director of the International Chair of Kinanthropometry, Universidad Católica San Antonio de Murcia
Other Study IDs: CE012109
Record Dates: First submitted 2021-05-24; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Body Weight; Body Fat Disorder
Keywords: Fat mass; Skinfolds; Anthropometry
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Caliper — Description of the sample adipose tissue and skinfolds using different calipers.

SUMMARY:
The present study aims to compare the results obtained from the assessment of skinfolds using four anthropometric calipers (Harpenden, Holtain, Slime Guide and Lipowise). The objectives are to check if there are differences depending on the caliper used to assess skinfolds, and to study the variation in skinfold compressibility as a function of the time elapsed from the application of the caliper to the measurement reading, as well as the validation of the Lipowise caliper. A cross-sectional study will be carried out with a sample of 100 university students aged between 18 and 25 years. Physical activity will be assessed by means of an International Physical Activity Questionnaire (IPAQ) and hydration status by urine samples. Anthropometric assessments, including weight, height, and eight skinfolds, will be performed according to the International Society for the Advancement in Kinanthropometry protocol, using the four previously mentioned calipers. Finally, a data analysis will be carried out to compare the results of the samples taken by the calipersand to draw conclusions.

DETAILED DESCRIPTION:
The objectives adressed in this study are: 1- To verify whether the model of adipometer used to measure skinfolds influences the results obtained. 2- To study the variation in skinfold compressibility as a function of the time elapsed between the application of the adipometer and the measurement reading.

To achieve the above objectives, it is proposed to carry out a ten-month cross-sectional study.

Sample:

The sample will consist of 80 university students (40 males and 40 females), caucasian, aged between 18 and 25 years. This is a convenience sample recruited in Spain.

The sample size was calculated based on previous criteria defined for validation studies, i.e. the number of subjects should be 7 times the number of items to be analysed and greater than or equal to 100. Taking into account that we will assess the 8 skinfolds defined by the International Society for the Advancement in Kinanthropometry (ISAK), and taking into account possible sample losses, should be recruited 50 participants of each sex.

Informed Consent All participants will be required to complete and sign the informed consent form, prior to the day of data collection, which we will designate as day 1, in a location that ensures their privacy, but in the presence of the investigator for clarification of any doubts that may arise. Participants will be reminded that: 1) their participation is voluntary and that they may leave the study if they wish; and 2) that all data collected are confidential.

Collection procedures

All assessments will be conducted on the same day, between 8:00 am and 2:00 pm, in a laboratory with a temperature of 24ºC and ambient humidity between 65-70%, and where participant privacy is guaranteed. Data collection from each participant will last an estimated 1 hour. On the day of data collection, participants must respect the following conditions:

* No physical exercise in the 12 hours prior to the evaluation, in the case of moderate exercise, or in the last 24 hours, in the case of vigorous exercise;
* Not to have consumed products with diuretic properties in the 24 hours prior to the assessment;
* Not having used a sauna in the 24 hours prior to the assessment;
* Not having a large meal the day before or on the day of the assessment;
* In the case of female participants, be between days 8 and 21 of the menstrual cycle.

Measurements Demographic data The following demographic data: date of birth, place/country of birth, sex, ethnicity, sporting practice (modality, level, years of practice, duration and weekly frequency of training) and day of the half cycle, will be obtained through a questionnaire. This questionnaire will be completed on the day the participant signs the informed consent form (day 1).

Physical Activity The assessment of physical activity will be carried out indirectly through the application of the IPAQ questionnaire - reduced version. This questionnaire shall be completed on day 1.

Hydration status Hydration status shall be assessed indirectly, using a urine colour scale. Immediately prior to the anthropometric assessment, the participant collects a portion of urine in a suitable container provided by the research team. In the presence of the participant, the urine will be graded according to its colour, after which it is discarded by the participant.

Anthropometric measurements All anthropometric measurements will be obtained by anthropometrists with current ISAK certification, respecting the procedures described by ISAK, always using the same measuring instruments. The assessments will begin with the measurement of height and body mass, using a Seca 217 portable stadiometer and a Seca 878 scale, respectively.

ELIGIBILITY:
Inclusion Criteria:

* To have signed the informed consent form
* To be a student of the San Antonio Catholic University of Murcia
* To be between 18 and 25 years old
* To have a BMI between 18.5 and 24.9
* Not have any metabolic or other disease that may affect body fat
* not have received hormonal or steroid treatment in the three months prior to the evaluation, with the exception of contraceptives.

Exclusion Criteria:

* To have indicators of changes in hydration status (signs of dehydration or oedema)
* To suffer an injury that compromises compliance with the ISAK assessment protocol.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population is conformed by students of different degrees. Finally, 102 students (46 males; 56 females) took part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Differences in anthropometry-estimated fat mass | Through study completion, an average of 10 months
  Analysis of the differences between the calipers, used in the same sample and with the same formulas

SECONDARY OUTCOMES:
Differences of the skinfolds sum | Through study completion, an average of 10 months
  Analysis of the differences between the calipers, used in the same sample and with the same formulas.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No